CLINICAL TRIAL: NCT04155658
Title: An in Situ Clinical Trial to Evaluate the Efficacy of a Calcium and Phosphate Enriched Sodium Monofluorophosphate Toothpaste on Enamel Lesion Remineralisation
Brief Title: Evaluation of Efficacy of Sodium Monofluorophosphate (SMPF) Toothpastes on Enamel Lesion Remineralisation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Collaborators: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: ORL-IST-3324
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Enamel Caries
MeSH Terms: interventions — Toothpastes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Experimental SMFP Toothpaste (Experimental): Toothpaste containing 1450ppm SMFP with additional calcium and phosphate
  Interventions: Other: Experimental Toothpaste containing 1450ppm SMFP
- SMFP Toothpaste (Active Comparator): Toothpaste containing 1450ppm SMFP
  Interventions: Other: Toothpaste containing 1450ppm SMFP
- Negative control toothpaste (Placebo Comparator): Toothpaste with no fluoride
  Interventions: Other: Toothpaste with no fluoride

INTERVENTIONS:
Other: Experimental Toothpaste containing 1450ppm SMFP — Experimental Toothpaste containing 1450ppm SMFP
  Arms: Experimental SMFP Toothpaste
Other: Toothpaste containing 1450ppm SMFP — Toothpaste containing 1450ppm SMFP
  Arms: SMFP Toothpaste
Other: Toothpaste with no fluoride — Toothpaste with no fluoride
  Arms: Negative control toothpaste

SUMMARY:
Double-blind, randomized, 3 group in situ study to assess effect of three toothpastes on enamel remineralization, as measured by change in integrated mineral loss (∆∆Z). The study will examine the efficacy of an experimental sodium monofluorophosphate (SMFP) toothpaste, a standard SMFP toothpaste and a negative control toothpaste with no fluoride.

DETAILED DESCRIPTION:
Double-blind, randomized, 3 group, in situ enamel remineralisation study. This study will accept up to 60 adult subjects who meet the inclusion/exclusion criteria in anticipation that at least 50 subjects will complete the study. All 60 subjects will have two human enamel specimens (one enamel specimen type C and one enamel specimen type N) placed in their partial denture for analysis by transverse microradiography (TMR) and of those sixty subjects, a subset will have an additional two enamel specimens (type N) placed in their partial denture for TMR measurement. All enamel specimens will have been partially demineralized using lactic acid in the laboratory prior to placement in subjects' dentures.

Subjects will receive a dental prophylaxis at the start of the trial and then brush their teeth with a fluoride-free toothpaste for the following 2 to 3 days. For the washout phase between each crossover period, subjects will return to brushing with their regular toothpaste for 4 to 5 days and then receive a dental prophylaxis and brush their teeth with a fluoride-free toothpaste for the 2 to 3 days before the next test period.

During each test period, subjects will be asked to brush with their allocated toothpaste at home twice daily for 4 weeks taking care to not brush the enamel specimens. The brushing procedure will be performed at home each morning following breakfast and right before going to bed on each evening. Subjects must wear their partial denture for 24 hours a day during the test phase.

At final visit of each test period, subjects will be instructed to brush their teeth with the randomly assigned trial toothpaste. Enamel specimens will be removed from denture and transferred to analyst for laboratory analyses.

ELIGIBILITY:
Key Inclusion Criteria:

1. Be wearing a removable mandibular partial denture that fits comfortably enough to wear 24 hours a day and willing to have their partial denture modified to accommodate the enamel test specimens.
2. Have completed and been accepted into the Oral Health Research Institute's screening for partial denture panel (#110007150).
3. Have no current active caries or periodontal disease that may compromise the trial or health of the person. Persons exhibiting localized periodontal conditions who, in the opinion of the trial dentist, will not be negatively affected by participation in intra-oral studies may be accepted. Persons with caries may participate if the carious lesions have been restored prior to beginning the first treatment.
4. Be willing to comply with all subjects' responsibilities (be willing and capable of wearing their removable partial dentures 24 hours per day during the treatment periods, attend appointments, follow brushing instructions, use non zinc adhesive in upper denture only etc.).
5. Have an unstimulated salivary flow rate of at least 0.2 ml per minute as determined by a five-minute salivary flow test at screening and a stimulated salivary flow rate of at least 0.8 ml per minute as determined by a two-minute stimulated (gum base) salivary flow test at screening

Key Exclusion Criteria:

1. Currently pregnant, intending to become pregnant during the trial period or breast-feeding.
2. Have a history of significant adverse effects following use of oral hygiene products such as toothpastes and mouth rinses.
3. Have any allergy to ingredients in the trial toothpaste products.
4. Currently be taking antibiotics or have taken antibiotics in the two weeks prior to the beginning the first treatment.
5. Have factors which could contraindicate their participation, such as any condition requiring the need for antibiotic premedication prior to a dental treatment, a condition requiring the need for long-term antibiotic use, blood thinning medications* that prohibit the safe conduct of a dental cleaning* or previous use of the weight loss medications Fen Phen® or Redux®. *Note: Subjects who are taking blood thinners in which written verification is obtained from their physician indicating their PT/INR levels (anti-coagulation blood levels) are at an acceptable level to avoid serious complications, such as bleeding during dental cleaning, may be accepted into the trial.
6. Currently taking or have ever taken a bisphosphonate drug (i.e. Fosamax®, Actonel®, Boniva®, Reclast®, or Zometa®) for treatment of osteoporosis.
7. Currently taking fluoride supplements, required to use a fluoride mouth rinse or have received a professional fluoride treatment in the two weeks preceding specimen placement.
8. Participation in another clinical trial/study within 30 days preceding the present trial/study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in integrated mineral loss from baseline ∆∆Z (enamel specimen type N) | Baseline to 4 weeks
  Calculation of Integrated Mineral Loss ∆Z = [(lesion depth x 87) - area under the curve] where 'area under the curve' relates volume % mineral at distances from the enamel specimen surface with respect to enamel section thickness, measured using transverse microradiography (TMR)

SECONDARY OUTCOMES:
Change in integrated mineral loss ∆∆Z (enamel specimen type C) | Baseline to 4 weeks
  Calculation of Integrated Mineral Loss ∆Z = [(lesion depth x 87) - area under the curve] where 'area under the curve' relates volume % mineral at distances from the enamel specimen surface with respect to enamel section thickness, measured using transverse microradiography (TMR)

CONTACTS AND LOCATIONS:
Overall Officials: Domenick T Zero, DDS, MS, Principal Investigator — Indiana University
Locations (1):
- Oral Health Research Institute, Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No